CLINICAL TRIAL: NCT04700423
Title: Efficacy and Safety of Moxidectin and Albendazole Compared to Ivermectin and Albendazole Co-administration in Adolescents Infected With Trichuris Trichiura: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of MOX/ALB vs. IVM/ALB Co-administration
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Public Health Laboratory Ivo de Carneri (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Dr., Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Moxi-ALB_IVM-ALB_combi-trial
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Trichuriasis; Ascariasis; Hookworm Infections; Helminthes; Infestation, Intestinal
Keywords: T. trichiura; A. lumbricoides; Hookworm; Soil-transmitted Helminths; Albendazole; Ivermectin; Moxidectin; Intestinal parasites; Anthelmintics
MeSH Terms: conditions — Trichuriasis; Ascariasis; Hookworm Infections; Helminthiasis; Ancylostomiasis; Intestinal Diseases, Parasitic | interventions — moxidectin; Albendazole; Ivermectin; Tablets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open Label with masked outcomes assessors
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- A: moxidectin (8 mg) / albendazole (400 mg) (Experimental): Combination therapy of moxidectin (8 mg using 2 mg tablets) plus albendazole (Zentel®, 400 mg, single tablet) administered orally at day 0
  Interventions: Drug: moxidectin (8 mg) / albendazole (400 mg)
- B: ivermectin (200 µg/kg) / albendazole (400 mg) (Active Comparator): Combination therapy of ivermectin (Stromectol®, 200 µg/kg using 3 mg tablets) plus albendazole (Zentel®, 400 mg, single tablet) administered orally at day 0
  Interventions: Drug: ivermectin (200 µg/kg) / albendazole (400 mg)
- C: albendazole (400 mg) (Active Comparator): Monotherapy of albendazole (400 mg) administered orally at day 0 Other names: Zentel®
  Interventions: Drug: ALBENDAZOLE 400 Mg ORAL TABLET [ZENTEL]
- D: ivermectin (200 µg/kg) (Active Comparator): Monotherapy of ivermectin ( 200 µg/kg using 3 mg tablets) administered orally at day 0 Other names: Stromectol®
  Interventions: Drug: ivermectin (200 µg/kg)
- E: moxidectin (8 mg) (Active Comparator): Monotherapy of moxidectin (8 mg using 2 mg tablets) administered orally at day 0
  Interventions: Drug: moxidectin (8 mg)

INTERVENTIONS:
Drug: moxidectin (8 mg) / albendazole (400 mg) — Combination therapy of moxidectin (8 mg using 2 mg tablets) plus albendazole (Zentel®, 400 mg, single tablet) administered orally at day 0
  Other Names: Zentel®
  Arms: A: moxidectin (8 mg) / albendazole (400 mg)
Drug: ivermectin (200 µg/kg) / albendazole (400 mg) — Combination therapy of ivermectin ((200 µg/kg), 3 mg tablet) plus albendazole (Zentel®, 400 mg, single tablet) administered orally at day 0
  Other Names: Stromectol® / Zentel®
  Arms: B: ivermectin (200 µg/kg) / albendazole (400 mg)
Drug: ALBENDAZOLE 400 Mg ORAL TABLET [ZENTEL] — Monotherapy of albendazole (Zentel®, 400 mg, single tablet) administered orally at day 0
  Other Names: Zentel®
  Arms: C: albendazole (400 mg)
Drug: ivermectin (200 µg/kg) — Monotherapy of ivermectin ((200 µg/kg), 3 mg tablet) administered orally at day 0
  Other Names: Stromectol®
  Arms: D: ivermectin (200 µg/kg)
Drug: moxidectin (8 mg) — Monotherapy of moxidectin (8 mg, using 2 mg tablets) administered orally at day 0
  Arms: E: moxidectin (8 mg)

SUMMARY:
The aim of this randomized controlled trial is to provide evidence on the efficacy and safety of co-administered moxidectin and albendazole compared to co-administered ivermectin and albendazole, and to assess the efficacy of the drug combinations compared to monotherapies in adolescents aged 12-19 years against infection with T. trichiura.

The efficacy of the different treatments will be determined 14-21 days, 5-6 weeks and 3 months post-treatment. Two fecal samples will be collected at each time-point assessment. The geometric mean based egg reduction rate (ERR) of T. trichiura egg counts will be assessed by Kato-Katz microscopy pre-treatment and 14-21 days post-treatment.

This trial will be conducted as a school-based study on Pemba Island (Zanzibar, Tanzania).

DETAILED DESCRIPTION:
We designed a non-inferiority trial to show that co-administered moxidectin and albendazole is non-inferior compared to co-administered ivermectin and albendazole in adolescents aged 12-19 years on Pemba Island (Tanzania). From previous studies conducted by our group, we expect similar efficacies from the combination moxidectin/ albendazole compared to ivermectin/ albendazole. However, moxidectin might be advantageous in terms of the drug's longer half-life and in areas with possible emerging ivermectin resistance. This study will allow comparing the efficacy of the two available co-administrations and will provide further insights on the potential value of moxidectin/ albendazole. Our data will pave the way for possible large scale, multi country follow-up studies. As recommended for new combination therapies, we simultaneously assess superiority of the drug combinations compared to monotherapies.

The primary objective is to demonstrate that co-administered moxidectin (8 mg) / albendazole (400 mg) is non-inferior to ivermectin (200 µg/kg) / albendazole (400 mg) in terms of egg reduction rates (ERRs) against T. trichiura infections assessed by Kato-Katz at 14-21 days post-treatment in adolescents aged 12-19 years using a non-inferiority margin of 2 percentage-points.

The secondary objectives of the trial are:

1. Efficacy assessments of combination therapies require demonstration of superiority against the respective monotherapies. Therefore, the trial has five different treatment groups: moxidectin (8 mg) / albendazole (400 mg) combination, ivermectin (200 µg/kg) / albendazole (400 mg) combination, albendazole (400 mg) monotherapy, ivermectin (200 µg/kg) monotherapy and moxidectin (8 mg) monotherapy.
2. to determine the CRs of the drug regimens against T. trichiura
3. to evaluate the safety and tolerability of the treatment
4. to determine the CRs and ERRs of the treatment schemes in study participants infected with hookworm and A. lumbricoides
5. to investigate potential extended effects on follow-up helminth prevalences (5-6 weeks and 3 months post-treatment) of the treatment regimens
6. to assess diagnostic performance and compare CRs based on egg counts retrieved from novel diagnostic tools (FECPAK-G2 and/or PCR) compared to standard microscopy
7. to characterize population PK parameters, as well as drug-drug interactions of active study treatments following single and co-administration in T. trichiura infected adolescents. If a dose-response is observed, a PK/PD analysis will further be performed

The study will be carried out in adolescents aged 12-19 years attending secondary schools on Pemba Island, Tanzania. After consenting, all participants will be asked to provide two stool samples (within a maximum of 7 days) at each time-point assesment. From each stool specimen, duplicate Kato-Katz thick smears (41.7 mg each) will be prepared and read under a microscope for eggs of T. trichiura, A. lumbricoides and hookworm by experienced technicians.

After randomization, all eligible adolescents will be treated with the respective single or combination treatment regimen according to their assigned treatment arm at day 0.

All drugs will be administered in the presence of the PI and/ co-PI, and ingestion confirmed. This will be recorded with the time and date of dosing. Participants will be kept for 3 hours after treatment administration to observe any possible acute AEs and reassessment will be done at 24h post-treatment. Additionally, interviews will be conducted to determine the emergence of clinical symptoms such as headache, abdominal pain, itching, nausea, vomiting and diarrhea directly before treatment within the scope of baseline assessment. At 3 and 24 hours after treatment and retrospectively at days 14 - 21 as well as 5-6 weeks and 3 months post-treatment, participants will again be interviewed for the assessment of adverse events (AEs).

Egg reduction rate calculated from the geometric means of co-administered moxidectin/ albendazole and ivermectin/ albendazole against T. trichiura assessed at 14-21 days post-treatment is the primary endpoint in our study.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 and 19 years.
* Written informed consent signed by either parents/caregivers for underage adolescents (aged 12-17 years) or by the participant him/herself (18-19 years of age); and written assent by underage participant.
* Agree to comply with study procedures, including provision of two stool samples at the beginning (baseline) and on three follow-up assessments (14-21 days, 5-6 weeks and 3 months after treatment).
* Willing to be examined by a study physician prior to treatment.
* At least two slides of the quadruple Kato-Katz thick smears positive for T. trichiura and infection intensities of at least 48 EPG.

Exclusion Criteria:

* No written informed consent by individual or caregiver and/or no written assent by minors
* Presence or signs of major systemic illnesses, e.g. body temperature ≥ 38°C, severe anemia (below 80g/l Hb according to WHO) upon initial clinical assessment.
* History of acute or severe chronic disease.
* Recent use of anthelmintic drug (within past 4 weeks).
* Attending other clinical trials during the study.
* Pregnancy, lactating, and/or planning to become pregnant within the next 6 months.
* Known allergy to study medications (i.e. albendazole, ivermectin or moxidectin).
* Taking medication with known interaction on study drugs.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 536 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Laboratory Ivo de Carneri, Chake Chake, Pemba, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Welsche S, Mrimi EC, Hattendorf J, Hurlimann E, Ali SM, Keiser J. Efficacy and safety of moxidectin and albendazole compared with ivermectin and albendazole coadministration in adolescents infected with Trichuris trichiura in Tanzania: an open-label, non-inferiority, randomised, controlled, phase 2/3 trial. Lancet Infect Dis. 2023 Mar;23(3):331-340. doi: 10.1016/S1473-3099(22)00589-8. Epub 2022 Oct 28. PMID 36354034
- [Derived] Welsche S, Mrimi EC, Keller L, Hurlimann E, Hofmann D, Hattendorf J, Ali SM, Keiser J. Efficacy and safety of moxidectin and albendazole compared to ivermectin and albendazole co-administration in adolescents infected with Trichuris trichiura: a randomized controlled trial protocol. Gates Open Res. 2021 Sep 27;5:106. doi: 10.12688/gatesopenres.13299.2. eCollection 2021. PMID 34632308

RESULTS

PARTICIPANT FLOW:
Period: Baseline/Treatment
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Started | 207 | 211 | 19 | 19 | 80
Completed | 207 | 211 | 19 | 19 | 80
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Follow-up 1: 14-21 Days Post Treatment
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Started | 207 | 211 | 19 | 19 | 80
Completed | 207 | 211 | 19 | 19 | 80
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Follow-up 2: 5-6 Weeks Post Treatment
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Started | 207 | 211 | 19 | 19 | 80
Completed | 206 | 211 | 18 | 19 | 80
Not Completed | 1 | 0 | 1 | 0 | 0
Period: Follow-up 3: 3 Months Post Treatment
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Started | 206 | 211 | 18 | 19 | 80
Completed | 201 | 210 | 18 | 18 | 77
Not Completed | 5 | 1 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg) | Total
Number analyzed (Participants) | 207 | 211 | 19 | 19 | 80 | 536
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (1.5) | 15.8 (1.5) | 15.6 (1.2) | 15.9 (1.3) | 15.8 (1.4) | 15.8 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 163 | 13 | 16 | 54 | 394
  Male | 59 | 48 | 6 | 3 | 26 | 142
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height, cm [Mean (Standard Deviation); unit: cm] | 157.1 (7.4) | 157.2 (7.3) | 159.1 (7.8) | 158.9 (7.1) | 157.4 (6.8) | 157.3 (7.3)
Weight, kg [Mean (Standard Deviation); unit: kg] | 48.3 (8.3) | 47.7 (8.2) | 50.8 (7.8) | 48.1 (6.1) | 47.1 (6.5) | 48.0 (7.9)
T. trichiura infection, geometric mean EPG [Geometric Mean (Standard Deviation); unit: eggs per gram] | 450 (4) | 468 (4) | 421 (4) | 573 (4) | 481 (3) | 463 (4)
T. trichiura infection, arithmetic mean EPG [Mean (Standard Deviation); unit: eggs per gram] | 975 (1329) | 1045 (1509) | 1014 (1504) | 1670 (3243) | 935 (1435) | 1022 (1525)
T. trichiura infection intensity (EPG): light [Count of Participants; unit: Participants] — T trichiura infection intensity categorised by mean EPG of stool (light 1-999, moderate 1000-9999, and heavy ≥10000)
  Eggs per gram (EPG) will be assessed by adding up the T. trichiura egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six.
  Participants | 144 | 148 | 14 | 14 | 57 | 377
T. trichiura infection intensity (EPG): moderate [Count of Participants; unit: Participants] — T trichiura infection intensity categorised by mean EPG of stool (light 1-999, moderate 1000-9999, and heavy ≥10000)
  Eggs per gram (EPG) will be assessed by adding up the T. trichiura egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six.
  Participants | 63 | 63 | 5 | 4 | 23 | 158
T. trichiura infection intensity (EPG): heavy [Count of Participants; unit: Participants] — T trichiura infection intensity categorised by mean EPG of stool (light 1-999, moderate 1000-9999, and heavy ≥10000)
  Eggs per gram (EPG) will be assessed by adding up the T. trichiura egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six.
  Participants | 0 | 0 | 0 | 1 | 0 | 1
Hookworm infection, No. infected [Count of Participants; unit: Participants] — Population: number of infected participants
  Participants | 64 | 70 | 3 | 8 | 28 | 173
Hookworm infection, geometric mean EPG [Geometric Mean (Standard Deviation); unit: eggs per gram] — Population: number of infected participants
  eggs per gram
    number analyzed (Participants) | 64 | 70 | 3 | 8 | 28 | 173
    (all) | 125 (4) | 112 (4) | 128 (8) | 94 (5) | 89 (3) | 111 (4)
Hookworm infection, arithmetic mean EPG [Mean (Standard Deviation); unit: eggs per gram] — Population: number of infected participants
  eggs per gram
    number analyzed (Participants) | 64 | 70 | 3 | 8 | 28 | 173
    (all) | 261 (332) | 261 (385) | 428 (644) | 200 (208) | 150 (175) | 243 (337)
Hookworm infection intensity (EPG): light [Count of Participants; unit: Participants] — Hookworm infection intensity is categorised by mean EPG of stool (light 1-1999, moderate 2000-3999, and heavy ≥4000).
  Eggs per gram (EPG) will be assessed by adding up the hookworm egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Population: Row population is the count of participants infected with Hookworm
  Participants
    number analyzed (Participants) | 64 | 70 | 3 | 8 | 28 | 173
    (all) | 64 | 70 | 3 | 8 | 28 | 173
A. lumbricoides infection, No. infected [Count of Participants; unit: Participants] | 106 | 110 | 12 | 14 | 50 | 292
A. lumbricoides infection, geometric mean EPG [Geometric Mean (Standard Deviation); unit: eggs per gram] — Population: number of infected participants
  eggs per gram
    number analyzed (Participants) | 106 | 110 | 12 | 14 | 50 | 292
    (all) | 7819 (4) | 5934 (5) | 8512 (4) | 4724 (4) | 6765 (4) | 6728 (4)
A. lumbricoides infection, arithmetic mean EPG [Mean (Standard Deviation); unit: eggs per gram] — Population: number of infected participants
  eggs per gram
    number analyzed (Participants) | 106 | 110 | 12 | 14 | 50 | 292
    (all) | 15823 (18844) | 14284 (20566) | 17062 (19533) | 9821 (9162) | 11969 (12883) | 14247 (18323)
A. lumbricoides intensity (EPG): light [Count of Participants; unit: Participants] — A lumbricoides infection intensity is categorised by mean EPG (light 1-4999, moderate 5000-49999, and heavy ≥50000).
  Eggs per gram (EPG) will be assessed by adding up the A. lumbricoides egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Population: Row population is the count of participants infected with A. lumbricoides
  Participants
    number analyzed (Participants) | 106 | 110 | 12 | 14 | 50 | 292
    (all) | 39 | 49 | 4 | 7 | 17 | 116
A. lumbricoides infection intensity (EPG): moderate [Count of Participants; unit: Participants] — A. lumbricoides infection intensity is categorised by mean EPG (light 1-4999, moderate 5000-49999, and heavy ≥50000).
  Eggs per gram (EPG) will be assessed by adding up the A. lumbricoides egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Population: Row population is the count of participants infected with A. lumbricoides
  Participants
    number analyzed (Participants) | 106 | 110 | 12 | 14 | 50 | 292
    (all) | 61 | 55 | 7 | 7 | 32 | 162
A. lumbricoides infection intensity (EPG): heavy [Count of Participants; unit: Participants] — A. lumbricoides infection intensity is categorised by mean EPG (light 1-4999, moderate 5000-49999, and heavy ≥50000).
  Eggs per gram (EPG) will be assessed by adding up the A. lumbricoides egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Population: Row population is the count of participants infected with A. lumbricoides
  Participants
    number analyzed (Participants) | 106 | 110 | 12 | 14 | 50 | 292
    (all) | 6 | 6 | 1 | 0 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Egg Reduction Rate Against T. Trichiura
Description: Egg reduction rate is calculated as the relative reduction in the group geometric mean egg output after co-administration of moxidectin/ albendazole and ivermectin/ albendazole assessed at 14-21 days post-treatment compared to the baseline levels.
Time Frame: 14-21 day post-treatment
Population: Geometric mean reduction in number of eggs at baseline and assessed at 14-21 days post-treatment
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 207 | 211 | 19 | 19 | 80
Percent change | 96.8 [95.8 to 97.6] | 99.0 [98.7 to 99.3] | 86.2 [61.8 to 95.6] | 94.2 [89.3 to 97.1] | 85.5 [79.7 to 89.8]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: The observation time for AE starts when the treatment is initiated. Subjects will be kept for observation for at least 3 hours following treatment for any acute AE and. If there is any abnormal finding, the local study physician will perform a full clinical examination and findings will be recorded. An emergency kit will be available on site to treat any medical conditions that warrant urgent medical intervention. Participants will also be interviewed at 3h and 24h as well as retrospectively 14 -21 days, 5-6 weeks and 3 months after treatment about the occurrence of AEs.
Time Frame: 3 hours, 24 hours, 14-21 days, 5-6 weeks and 3 months post-treatment
Population: number analyzed corresponds to the number of participants assessed per time point
Measure: Count of Participants; unit: Participants
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 207 | 211 | 19 | 19 | 80
Participants
  Baseline | 7 | 9 | 0 | 0 | 0
  3h post treatment | 17 | 25 | 0 | 2 | 6
  24h post treatment: number analyzed (Participants) | 205 | 211 | 19 | 19 | 80
  24h post treatment | 36 | 40 | 3 | 2 | 6
  14 to 21 days post treatment | 35 | 41 | 4 | 4 | 13
  5 to 6 weeks post treatment: number analyzed (Participants) | 206 | 211 | 18 | 19 | 80
  5 to 6 weeks post treatment | 20 | 10 | 2 | 2 | 6
  3 months post treatment: number analyzed (Participants) | 201 | 210 | 18 | 18 | 77
  3 months post treatment | 10 | 15 | 0 | 2 | 4

3. Secondary Outcome: Superiority in Terms of Cure Rates (CRs)
Description: Assessment of superiority in terms of CRs of the drug combinations compared to their corresponding monotherapies: Arm C: Albendazole (400 mg) Arm D: Ivermectin (200 μg/kg) and Arm E: Moxidectin (8 mg). Cure rates is defined as the percentages of participants treated with Moxidectin (8 mg)/Albendazole (400 mg), Ivermectin (200 μg/kg)/Albendazole (400 mg), Albendazole (400 mg), Ivermectin (200 μg/kg) or Moxidectin (8 mg) who were cured of infections with T. trichiura.
Time Frame: 14-21 day post-treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 207 | 211 | 19 | 19 | 80
Percentage of participants | 34.3 [27.9 to 41.2] | 54.0 [47.1 to 60.9] | 26.3 [9.1 to 51.2] | 10.5 [1.3 to 33.1] | 11.2 [5.3 to 20.3]

4. Secondary Outcome: Cure Rates Against T. Trichiura
Description: Cure rates of each treatment will be calculated as the percentage of egg-positive participants at baseline who become egg-negative after treatment.
Time Frame: 14-21 day post-treatment
Population: Number of participants found positive for hookworm at 14-21 days post-treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 207 | 211 | 19 | 19 | 80
Percentage of participants | 34.3 [27.9 to 41.2] | 54.0 [47.1 to 60.9] | 26.3 [9.1 to 51.2] | 10.5 [1.3 to 33.1] | 11.2 [5.3 to 20.3]

5. Secondary Outcome: Extended Effects (Egg Reduction Rate) on Follow-up of T. Trichiura: 5-6 Weeks
Description: Eggs per gram of stool will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the two treatment arms before and after treatment to assess the corresponding ERRs.
Time Frame: 5-6 weeks post-treatment
Population: Geometric mean reduction in number of eggs at baseline and assessed at 5-6 weeks post-treatment
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 206 | 211 | 18 | 19 | 80
Percent change | 97.0 [96.0 to 97.8] | 98.3 [97.6 to 98.7] | 75.7 [40.8 to 90.5] | 76.9 [65.6 to 84.7] | 85.4 [77.6 to 90.7]

6. Secondary Outcome: Extended Effects (Cure Rate) on Follow-up of T. Trichiura: 5-6 Weeks
Description: as for outcome 4
Time Frame: 5-6 weeks post-treatment
Population: Number of participants found positive for hookworm at 5-6 weeks post-treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 206 | 211 | 18 | 19 | 80
Percentage of participants | 37.4 [30.8 to 44.4] | 46.4 [39.6 to 53.4] | 16.7 [3.6 to 41.4] | 0.0 [0.0 to 17.6] | 11.2 [5.3 to 20.3]

7. Secondary Outcome: Extended Effects (Egg Reduction Rate) on Follow-up of T. Trichiura: 3 Months
Description: as for outcome 5
Time Frame: 3 months post-treatment
Population: Geometric mean reduction in number of eggs at baseline and assessed at 3 months post-treatment
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 201 | 210 | 18 | 18 | 77
Percent change | 93.2 [90.8 to 95.0] | 97.1 [96.1 to 97.9] | 78.2 [55.5 to 90.0] | 55.4 [22.3 to 74.2] | 71.9 [58.9 to 81.4]

8. Secondary Outcome: Extended Effects (Cure Rates) on Follow-up of T. Trichiura: 3 Months
Description: as for outcome 4
Time Frame: 3 months post-treatment
Population: Number of participants found positive for T. trichiura at baseline and assessed at 3 months post-treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 201 | 210 | 18 | 18 | 77
Percentage of participants | 27.4 [21.3 to 34.1] | 39.5 [32.9 to 46.5] | 11.1 [1.4 to 34.7] | 0.0 [0.0 to 18.5] | 9.1 [3.7 to 17.8]

9. Secondary Outcome: Egg Reduction Rates Against Concomitant Soil-transmitted Helminth Infections: Hookworm
Description: as for outcome 5
Time Frame: 14-21 days post-treatment
Population: Geometric mean reduction in number of eggs at baseline and assessed at 14-21 days post-treatment
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 64 | 70 | 3 | 8 | 28
Percent change | 98.8 [97.6 to 99.4] | 97.4 [95.9 to 98.4] | 100.0 [100.0 to 100.0] | 61.9 [-8.0 to 86.8] | 81.2 [58.9 to 91.7]

10. Secondary Outcome: Cure Rates Against Concomitant Soil-transmitted Helminth Infections: Hookworm
Description: as for outcome 4
Time Frame: 14-21 days post-treatment
Population: Number of participants found positive for hookworm at baseline and assessed at 14-21 days post-treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 64 | 70 | 3 | 8 | 28
Percentage of participants | 75.0 [62.6 to 85.0] | 62.9 [50.5 to 74.1] | 100.0 [29.2 to 100.0] | 25.0 [3.2 to 65.1] | 32.1 [15.9 to 52.4]

11. Secondary Outcome: Extended Effects (Egg Reduction Rate) on Follow-up of Hookworm: 5-6 Weeks
Description: as for outcome 5
Time Frame: 5-6 weeks post-treatment
Population: Mean number of participants found positive for hookworm at 5-6 weeks post-treatment
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 64 | 70 | 3 | 8 | 28
Percent change | 98.6 [97.4 to 99.3] | 96.8 [94.9 to 98.1] | 94.6 [56.9 to 100.0] | 57.9 [-10.4 to 84.3] | 88.7 [71.0 to 95.9]

12. Secondary Outcome: Extended Effects (Cure Rate) on Follow-up of Hookworm: 5-6 Weeks
Description: as for outcome 4
Time Frame: 5-6 weeks post-treatment
Population: Number of participants found positive for hookworm at 5-6 weeks post-treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 64 | 70 | 3 | 8 | 28
Percentage of participants | 71.9 [59.2 to 82.4] | 61.4 [49.0 to 72.8] | 66.7 [9.4 to 99.2] | 25.0 [3.2 to 65.1] | 42.9 [24.5 to 62.8]

13. Secondary Outcome: Extended Effects (Egg Reduction Rate) on Follow-up of Hookworm: 3 Months
Description: as for outcome 5
Time Frame: 3 months post-treatment
Population: Geometric mean reduction in number of eggs at baseline and assessed at 3 months post-treatment
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 62 | 70 | 3 | 8 | 25
Percent change | 97.6 [95.9 to 98.7] | 95.1 [91.5 to 97.3] | 96.3 [83.6 to 100.0] | 56.1 [-31.9 to 85.5] | 76.7 [39.3 to 92.0]

14. Secondary Outcome: Extended Effects (Cure Rate) on Follow-up of Hookworm: 3 Months
Description: as for outcome 4
Time Frame: 3 months post-treatment
Population: Number of participants found positive for hookworm at 3 months post-treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 62 | 70 | 3 | 8 | 25
Percentage of participants | 66.1 [53.0 to 77.7] | 60.0 [47.6 to 71.5] | 66.7 [9.4 to 99.2] | 25.0 [3.2 to 65.1] | 32.0 [14.9 to 53.5]

15. Secondary Outcome: Egg Reduction Rates Against Concomitant Soil-transmitted Helminth Infections: Ascaris Lumbricoides
Description: Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the two treatment arms before and after treatment to assess the corresponding ERRs.
Time Frame: 14-21 days post-treatment
Population: Geometric mean reduction in number of eggs at baseline and assessed at 14-21 days post-treatment
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 106 | 110 | 12 | 14 | 50
Percent change | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

16. Secondary Outcome: Cure Rates Against Concomitant Soil-transmitted Helminth Infections: Ascaris Lumbricoides
Description: Cure rates is defined as the percentages of participants treated with Moxidectin (8 mg)/Albendazole (400 mg), Ivermectin (200 μg/kg)/Albendazole (400 mg), Albendazole (400 mg), Ivermectin (200 μg/kg) or Moxidectin (8 mg) who were cured of infections with A. lumbricoides.
Time Frame: 14-21 days post-treatment
Population: Number of participants found positive for A. lumbricoides at baseline and assessed at 14-21 days post-treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 106 | 110 | 12 | 14 | 50
Percentage of participants | 100.0 [96.6 to 100.0] | 96.4 [91.0 to 99.0] | 91.7 [61.5 to 99.8] | 100.0 [76.8 to 100.0] | 98.0 [89.4 to 99.9]

17. Secondary Outcome: Extended Effects (Egg Reduction Rate) on Follow-up of A. Lumbricoides: 5-6 Weeks
Description: as for outcome 5
Time Frame: 5-6 weeks post-treatment
Population: Geometric mean reduction in number of eggs at baseline and assessed at 5-6 weeks post-treatment
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 106 | 110 | 12 | 14 | 50
Percent change | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

18. Secondary Outcome: Extended Effects (Cure Rate) on Follow-up of A. Lumbricoides: 5-6 Weeks
Description: as for outcome 4
Time Frame: 5-6 weeks post-treatment
Population: Number of participants found positive for hookworm at 5-6 weeks post-treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 106 | 110 | 12 | 14 | 50
Percentage of participants | 100.0 [100.00 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 98.0 [89.4 to 99.9]

19. Secondary Outcome: Extended Effects (Egg Reduction Rate) on Follow-up of A. Lumbricoides: 3 Months
Description: as for outcome 5
Time Frame: 3 months post-treatment
Population: Geometric mean reduction in number of eggs at baseline and assessed at 3 months post-treatment
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 102 | 110 | 12 | 14 | 48
Percent change | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [99.9 to 100.0] | 100.0 [99.9 to 100.0] | 100.0 [99.9 to 100.0]

20. Secondary Outcome: Extended Effects (Cure Rate) on Follow-up of A. Lumbricoides: 3 Months
Description: as for outcome 4
Time Frame: 3 months post-treatment
Population: Number of participants found positive for hookworm at 3 months post-treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
Number analyzed (Participants) | 102 | 110 | 12 | 14 | 48
Percentage of participants | 87.3 [79.2 to 93.0] | 88.2 [80.6 to 93.6] | 91.7 [61.5 to 99.8] | 92.9 [66.1 to 99.8] | 87.5 [74.8 to 95.3]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed 3h and 24h post-treatment. At the three follow-up timepoints of 14-21 days, 5-6 weeks, and 3 months after treatment, adverse events were assessed retrospectively
Description: Severity grading was categorized according to the US National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE; version 5.0)
Arm/Group | A: Moxidectin (8 mg) / Albendazole (400 mg) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) | C: Albendazole (400 mg) | D: Ivermectin (200 µg/kg) | E: Moxidectin (8 mg)
All-Cause Mortality (participants affected / at risk) | 0/207 | 0/211 | 0/19 | 0/19 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/207 | 0/211 | 0/19 | 0/19 | 0/80
Other Adverse Events (participants affected / at risk) | 73/207 | 93/211 | 4/19 | 6/19 | 23/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Moxidectin (8 mg) / Albendazole (400 mg) (N=207) | B: Ivermectin (200 µg/kg) / Albendazole (400 mg) (N=211) | C: Albendazole (400 mg) (N=19) | D: Ivermectin (200 µg/kg) (N=19) | E: Moxidectin (8 mg) (N=80)
Headache (General disorders) | 30 | 38 | 3 | 2 | 6
Abdominal pain (General disorders) | 13 | 16 | 1 | 1 | 4
Itching (General disorders) | 4 | 8 | 0 | 1 | 1
Dizziness (General disorders) | 1 | 3 | 0 | 0 | 1
Musculoskeletal pain (General disorders) | 6 | 6 | 0 | 1 | 3
Muscle weakness (General disorders) | 6 | 9 | 0 | 0 | 4
Rash (General disorders) | 2 | 4 | 0 | 1 | 0
Nausea (General disorders) | 3 | 3 | 0 | 0 | 1
Diarrhea (General disorders) | 1 | 5 | 0 | 0 | 1
Cough (General disorders) | 0 | 0 | 0 | 0 | 0
Constipation (General disorders) | 3 | 1 | 0 | 0 | 0
Vomiting (General disorders) | 1 | 0 | 0 | 0 | 2
Other (General disorders) | 3 | 0 | 0 | 0 | 0 — Adverse events assessment of self-reported fever, sleepiness, itching eyes, eye discharge, flu-like symptoms, ear pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT04700423/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT04700423/ICF_001.pdf